CLINICAL TRIAL: NCT00910910
Title: A Phase 3, Multicenter, Randomized, Openlabel, Parallel-Group Study of the Efficacy and Safety of Lenalidomide (Revlimid®) Versus Chlorambucil as First-Line Therapy for Previously Untreated Elderly Patients With B-Cell Chronic Lymphocytic Leukemia (The Origin Trial)
Brief Title: Study Of The Effectiveness & Safety Of Lenalidomide Versus Chlorambucil As First Line Therapy For Elderly Patients With B-Cell CLL (The ORIGIN Trial)
Acronym: ORIGIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-CLL-008; 2008-003079-32 (EudraCT Number)
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Lenalidomide (Experimental): 1 - Lenalidomide
  Interventions: Drug: Lenalidomide
- 2- Chlorambucil (Active Comparator): 2- Chlorambucil
  Interventions: Drug: Chlorambucil

INTERVENTIONS:
Drug: Lenalidomide — For patients with normal renal function (defined as CrCl ≥ 60 mL/min), 5 mg once daily on Days 1 through 28 of the first 28-day cycle, 10 mg once daily on Days 1 through 28 starting at the second cycle, 15 mg once daily starting at the third cycle and for the remainder of the study until PD or unacceptable toxicity, whichever occurs first.
  For patients with moderate renal impairment (defined as CrCl ≥ 30 to < 60 mL/min), 2.5 mg once daily on Days 1 through 28 of the first 28-day cycle, 5 mg once daily on Days 1 through 28 starting at the second cycle, 7.5 mg once daily starting at the third cycle and for the remainder of the study until PD or unacceptable toxicity, whichever occurs first.
  Other Names: Revlimid
  Arms: 1 - Lenalidomide
Drug: Chlorambucil — Patients assigned to the chlorambucil arm will receive oral chlorambucil tablets at 0.8 mg/kg on Days 1 and 15 of each 28-day cycle for a total duration of 12 months (approximately 13 cycles).
  Other Names: Leukeran
  Arms: 2- Chlorambucil

SUMMARY:
The purpose of this study is to determine the safety and efficacy of lenalidomide as a first line therapy in treating patients with B-cell Chronic Lymphocytic Leukemia. This study will compare the effects (good and bad) of lenalidomide with chlorambucil.

DETAILED DESCRIPTION:
After notification from the US Food and Drug Administration (FDA) on 12 July 2013, Celgene agreed to discontinue the lenalidomide treatment for all patients due to an imbalance in the number of deaths in patients treated with lenalidomide versus patients treated with chlorambucil. No specific causality for this imbalance has been identified to date. Investigators were instructed to immediately discontinue all participants from experimental lenalidomide treatment and inform their patients accordingly. Participants on the Chlorambucil arm may continue up to 12 months (13 cycles) with the last participant completing in March 2014. All randomized participants will continue to be followed for overall survival and secondary primary malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an informed consent form.
2. Age ≥ 65 years
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Must have a documented diagnosis of B-cell CLL.
5. Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.
6. Must agree to follow pregnancy precautions as required by the protocol.
7. Must agree to receive counseling related to teratogenic and other risks of lenalidomide.
8. Must agree not to donate blood or semen as defined by the protocol

Exclusion Criteria:

1. Prior treatment for B-cell CLL.
2. Any medical condition, that would prevent the subject from signing the informed consent form.
3. Active infections requiring systemic antibiotics.
4. Systemic infection that has not resolved > 2 months prior to initiating lenalidomide
5. Pregnant or lactating females.
6. Participation in any clinical study or having taken any investigational therapy within 28 days.
7. Known presence of alcohol and/or drug abuse.
8. Central nervous system (CNS) involvement.
9. Prior history of malignancies, other than CLL, unless the subject has been free of the disease for ≥3 years. Exceptions include the following:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
10. History of renal failure requiring dialysis.
11. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection.
12. Prior therapy with lenalidomide.
13. Evidence of TLS at screening
14. Presence of specific hematology and/or chemistry abnormalities
15. Uncontrolled hyperthyroidism or hypothyroidism
16. Venous thromboembolism within one year
17. ≥ Grade-2 neuropathy
18. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
19. Disease transformation [i.e. Richter's Syndrome (lymphomas) or prolymphocytic leukemia]

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-10-13 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jones, MD, Study Director — Celgene Corporation
Locations (165):
- United States (28):
  - California Cancer Associates for Research and Excellence cCARE, Escondido, California
  - Innovative Clinical Research Institute, Whittier, California
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - University Hematology Oncology Inc., Centralia, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Medical Consultants, PC, Muncie, Indiana
  - Floyd Memorial Cancer Center of Indiana, a division of Floyd Memorial Hospital and Health Services, New Albany, Indiana
  - Purchase Cancer Group, Paducah, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Oncology and Hematology Associates, PA, Denville, New Jersey
  - The Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Somerset Hematology-Oncology Associates, Somerville, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Drexel University, College of Medicine, Philadelphia, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Berks Hematology-Oncology Associates, West Reading, Pennsylvania
  - Geisinger Health System, Wilkes-Barre, Pennsylvania
  - Charleston Hematology Oncology P.A., Charleston, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Central Texas Veterans Health Care System, Temple, Texas
  - Swedish Tumor Institute, Seattle, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - Columbia St Marys Cancer Center, Milwaukee, Wisconsin
- Australia (9):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - IMVS, Adelaide, South Australia
  - Western Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Flinders Medical Centre, Bedford Park
  - St. Vincent Hospital, Fitzroy
  - Nepean Hospital, Kingswood, NSW
  - Calvary Mater Hospital, Waratah
  - Westmead Hospital Australia, Westmead
- Austria (2):
  - Universitaetsklinik Innsbruck, Innsbruck
  - Medical University of Vienna Internalmedicine 1, Hematology, Vienna
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Hopital Erasme, Brussels
  - Hopital de Jolimont, Haine-Saint-Paul
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU Mont -Godinne, Yvoir
- Brazil (14):
  - Monte Tabor - Hospital Sao Rafael, Salvador, Estado de Bahia
  - BIOCANCER - Centro de Pesquisa e Tratamento do Câncer S/A, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Universitario de Brasilia, Brasílía
  - Hospital Erasto Gaertner, Curitiba
  - Pro Onco Centro de Tratamento Oncologico, Londrina
  - Hospital Israelita Albert Einstein, Morumbi
  - Instituto Estadual Arthur de Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Instituto Nacional de Cancer - INCA, Rio de Janeiro
  - Centro de Estudos e Pesquisas de Hematologia e Oncologia da Faculdade de Medicina do ABC, Santo André
  - Instituto de Ensino e Pesquisa Sao Lucas, São Paulo
  - Fundação Antonio Prudente - AC Camargo Câncer center, São Paulo
- Bulgaria (5):
  - MHAT Georgi Stranski PlevenHematology Clinic, Pleven
  - University hospital Sveti Georgi Hematology Clinic, Plovdiv
  - Military Medical Academy, Sofia
  - National Specialized Hospital for Active Treatment of Hematology Diseases, Sofia
  - University hospital Sveta Marina, Varna
- Canada (4):
  - Regional Health Authority B-Saint John Regional Hospital, Saint John, New Brunswick
  - General Hospital, Eastern Health, St. John's, Newfoundland and Labrador
  - Hospital Charles LeMoyne, Greenfield Park, Quebec
  - Sacre-Couer Hospital, Montreal, Quebec
- Chile (2):
  - Instituto Oncologico, Reñaca
  - Instituto Clinico Oncologico del Sur ICOS, Temuco
- Oncomedica S.A., Montería, Colombia
- Croatia (4):
  - University Hospital Centre Split, Split
  - General Hospital Sveti Duh, Zagreb
  - Klinicka bolnica Dubrava Klinika za unutarnje bolesti Odjel za Hematologiju, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (3):
  - University Hospital2.Dep.Intern.Med. Hematology, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Faculty Hospital Kralovske Vinohrady, Prague
- Denmark (3):
  - Rigshospitalet University Hospital, Copenhagen
  - Herlev University Hospital Dep of hematology, Harlev
  - Roskilde University Hospital, Roskilde
- France (6):
  - Bergonie Institut, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHRU, Grenoble
  - CHU Dupuytren, Limoges
  - Hopital de l'Archet 1, Nice
  - CHU Hautepierre, Strasbourg
- Hungary (5):
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Kaposi Mor Oktato Korhaz, Kaposvár
  - Szegedi TudomanyegyetemII Belgyogyaszati Klinika, Szeged
  - Komarom-Esztergom Megye Onkormanyzat Szent Borbala Korhaza, Tatabánya
  - Petz Aladar Country Hospital, Vasvari Pal U. 2
- Israel (11):
  - Ha'Emek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Bnei Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center Department of Hematology, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (14):
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCSS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Ospedale San Raffaele S.r.l., Milan
  - Istituto Europeo di Oncologia - IEO, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Ospedale Cardarelli, Naples
  - Universita del Piemonte Orientale, Novara
  - AOU San Luigi Gonzaga, Orbassano
  - Universita degli Studi di Padova, Padua
  - Ospedale S. Chiara, Pisa
  - Azienda Ospedaliera Ospedale San Carlo, Potenza
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - Ospedale Umberto I, Torrette Di Ancona
- Netherlands (3):
  - Maxima Medisch Centrum, Eindhoven
  - Spaame Ziekenhuis, Hoofddorp
  - Isala Klinieken, Zwolle
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - North Shore University Hospital, Takapuna
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewodzki Szpital Specjalistczny im. Mikolaja Kopernika, Lodz
  - Specjalistyczny Szpital miejski im. Kopernika, Torun
  - Klinika Chorob wewnetrznych i Hematologii, Warsaw
  - Nowotworww Krwi i Transplantacji Szpiku, Wroclaw
- Portugal (2):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Portugues Oncologia do Porto Francisco Gentil EPE, Porto
- Romania (5):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf Spiridon Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (11):
  - Archangelsk Regional Clinical Hospital, Arkhangelsk
  - City Hospital 8, Barnaul
  - Russian Academy of Medical Sciences Institution, Moscow
  - Moscow GUZ City Clinical Hospital, Moscow
  - NUZ Central Clinical Hospital, Moscow
  - GUZ Nizhegorodskaya Regional Clinical Hospital, Nizhny Novgorod
  - MUZ City clinical hospital, Novosibirsk
  - St. Petersburg Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - GUS Leningrad Regional Clinical Hospital, Saint Petersburg
  - Federal Centre of Heart, Blood and Endocrinology of Rosmed technlologies V.A. Almazov, Saint Petersburg
  - Regional Clinical Hospital 1, Yekaterinburg
- Serbia (2):
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - Martinska Fakultna Nemocnica, Martin
- South Africa (3):
  - University Witwatersrand Oncology, Parktown
  - Pretoria Academic Hospital, Pretoria
  - Mary Potter Oncology Centre, Pretoria
- Spain (10):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitario Vall D hebron, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda
  - Hospital General Universitario Morales Messeguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario La Fe, Valencia
- United Kingdom (3):
  - Royal Bournemouth General Hospital, Bournemouth
  - St. Bartholomew's and The Royal London Hospital, London
  - St George's Healthcare NHS Trust, London

REFERENCES:
- [Result] Chanan-Khan A, Egyed M, Robak T, Martinelli de Oliveira FA, Echeveste MA, Dolan S, Desjardins P, Blonski JZ, Mei J, Golany N, Zhang J, Gribben JG. Randomized phase 3 study of lenalidomide versus chlorambucil as first-line therapy for older patients with chronic lymphocytic leukemia (the ORIGIN trial). Leukemia. 2017 May;31(5):1240-1243. doi: 10.1038/leu.2017.47. Epub 2017 Jan 31. No abstract available. PMID 28140392
- See also: Related Info — https://www.nature.com/articles/leu201747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 118 sites randomized participants in Austria, Australia, Belgium, Brazil, Bulgaria, Canada, Chile, Columbia, Croatia, Czech Republic, Denmark, Hungary, Israel, Italy, the Netherlands, New Zealand, Poland, Portugal, Romania, Russia, South Africa, Slovakia, Spain, Serbia, the United Kingdom, and the United States of America
Pre-assignment Details: Participants were randomized 1:1 to lenalidomide or chlorambucil and stratified by disease stage, presence of pre-defined co-morbidities and presence of at least one of the following poor prognostic factors: 11q deletion, 17 p deletion, unmutated IgVH and B2M>4.0 mg/dL.
Groups:
- Lenalidomide: For participants with normal renal function [defined as Creatinine Clearance (CrCL ) ≥ 60 mL/min], 5 mg lenalidomide by mouth (PO) once daily (QD) on Days 1 through 28 of the first 28-day cycle, 10 mg lenalidomide PO QD on Days 1 through 28 starting at cycle 2, 15 mg lenalidomide PO QD starting at cycle 3 and for the remainder of the study until progressive disease (PD) or unacceptable toxicity, whichever occurred first. For participants with moderate renal impairment (defined as CrCL ≥ 30 to < 60 mL/min), 2.5 mg lenalidomide PO QD on Days 1 through 28 of the first 28-day cycle, 5 mg lenalidomide PO QD on Days 1 through 28 starting at cycle 2, 7.5 mg lenalidomide PO QD starting at cycle 3 and for the remainder of the study until PD or unacceptable toxicity, whichever occurred first.
- Chlorambucil: Chlorambucil oral tablets at 0.8 mg/kg on Days 1 and 15 of each 28-day cycle for a total duration of 12 months (approximately 13 cycles).
Period: Overall Study
Arm/Group | Lenalidomide | Chlorambucil
Started | 225 | 225
Safety Population | 224 (All randomized participants who received at least 1 dose of the either lenalidomide or chlorambucil) | 223 (All randomized participants who received at least 1 dose of the either lenalidomide or chlorambucil)
Completed | 0 (Completed includes participants who continued with ongoing treatment) | 1 (Completed includes participants who continued with ongoing treatment)
Not Completed | 225 | 224
Not completed — Adverse Event | 63 | 35
Not completed — PD without histologic change | 27 | 23
Not completed — PD with histologic change | 0 | 2
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 9 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Completed 13 cycles of treatment | 0 | 118
Not completed — Other | 114 | 32
Not completed — Untreated before cycle 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was defined as all participants who were randomized, independent of whether they received study treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Chlorambucil | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (5.72) | 73.3 (5.72) | 73.1 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants] — The Intent-to-Treat (ITT) population was defined as all participants who were randomized, independent of whether they received study treatment or not.
  Participants
    Female | 93 | 83 | 176
    Male | 132 | 142 | 274

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to the first documented progression confirmed per investigator's assessment or death due to any cause on study, whichever occurred first. The progression date was assigned to the earliest time when any progression was observed without prior missing assessments. If withdrawal of consent or lost to follow-up occurred before documented progression or death, then these observations were censored at the date when the last complete tumor assessments determined a lack of progression
Time Frame: From first dose of study drug to date of data cut-off of 18 Feb 2013; up to approximately 39 months
Population: This is a smaller population used in this analysis (earlier cut-off date) prior to the last participant enrolled in the study. The ITT population was defined as all participants who were randomized, independent of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 212 | 215
months | 30.8 [18.7 to NA] — Not Applicable = The upper boundary of confidence interval (CI) is not estimable because of censored participants. | 23.0 [19.3 to 29.2]
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Stratification factors: Disease stage (Binet A or Binet B or Rai I or Rai II versus (VS) Binet C or Rai III or Rai IV); Presence of at least one of the co-morbidities Asparate transaminase (AST)/Alanine transaminase (ALT) ≥ 3.0 times Upper Limits of Normal (ULN,) Creatinine clearance ≥ 30 to < 60 mL/min, Yes VS No); Presence of at least one 11q deletion, 17p deletion, unmutated Immunoglobulin Heavy-chain Variable-region (IgVH) or Beta-2 Microglobulin (ß2M )> 4.0 mg/L (Yes versus No VS Unknown); Test type: Superiority; p = 0.323, stratified log rank; Hazard Ratio (HR) = 1.21, 90% CI 2-sided [0.88 to 1.66] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

2. Primary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS) With a Later Cut-off Date of 14 March 2014
Description: Progression-free survival was defined as the time from randomization to the first documented progression confirmed per investigator's assessment or death due to any cause on study, whichever occurred first. Progressive disease included lymphadenopathy, an appearance of any new lesion such as enlarged lymph nodes (> 1.5 cm), splenomegaly, hepatomegaly or other organ infiltrates, an increase by 50% or more in greatest determined diameter of any previous site or an increase by 50% or more in the sum of the product of diameters of multiple nodes. The progression date was assigned to the earliest time when any progression was observed without prior missing assessments. If withdrawal of consent or lost to follow-up occurred before documented progression or death, then these observations were censored at the date when the last complete tumor assessments determined a lack of progression.
Time Frame: From randomization to data cut off date of 31 March 2014; median follow up time for all participants was 12.6 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 225 | 225
months | 30.8 [18.7 to NA] — NA = The upper boundary of CI is not estimable because of censored participants. | 21.4 [19.3 to 25.1]
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.967, Log Rank — The p-value is based on a stratified log-rank test; Cox Proportional Hazard = 0.99, 90% CI 2-sided [0.76 to 1.29] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs = any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, regardless of cause. Serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs were graded based upon the participants symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0); AEs were evaluated for severity according to the following scale: Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death
Time Frame: From randomization up to data cut-off of 18 Feb 2013; Up to approximately 39 months; maximum duration of exposure for Lenalidomide was 1086 days and 406 days for Chlorambucil
Population: This is a smaller population used in this analysis (earlier cut-off date) prior to the last participant enrolled in the study. The safety population was defined as all randomized participants who received at least 1 dose of the study treatment (either lenalidomide or chlorambucil) as of the data cut off date of 18 Feb 2013
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 211 | 213
participants
  ≥ 1 TEAE | 202 | 186
  ≥ 1 TEAE related to study drug | 183 | 139
  ≥ 1 NCI CTC Grade 3-4 TEAE | 173 | 117
  Grade 3-4 adverse event related to any study drug | 143 | 82
  ≥ 1 NCI CTC Grade 5 TEAE | 21 | 9
  ≥ Grade 5 adverse event related to any study drug | 6 | 1
  ≥ 1 Serious TEAE | 129 | 76
  ≥ 1 Serious TEAE related to any study drug | 95 | 46
  ≥1 TEAE leading to stopping either study drug | 61 | 34
  ≥1 Related TEAE leading to stopping either drug | 39 | 19

4. Secondary Outcome: Number of Participants With Adverse Events With a Later Cut-off Date of 31 March 2014
Description: as for outcome 3
Time Frame: From randomization to the data cut-off date of 31 March 2014; Up to 53 months; maximum duration of exposure for Lenalidomide was 1140 days and 406 days for Chlorambucil
Population: The safety population was defined as all randomized participants who received at least 1 dose of the study treatment (either lenalidomide or chlorambucil).
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 224 | 223
participants
  ≥ 1 TEAE | 216 | 202
  ≥ 1 TEAE related to study drug | 194 | 155
  ≥ 1 NCI CTC Grade 3-4 TEAE | 188 | 131
  Grade 3-4 adverse event related to any study drug | 157 | 90
  ≥ 1 NCI CTC Grade 5 TEAE | 21 | 11
  ≥ Grade 5 adverse event related to any study drug | 6 | 1
  ≥ 1 Serious TEAE | 148 | 90
  ≥ 1 Serious TEAE related to any study drug | 107 | 53
  ≥1 TEAE leading to stopping either study drug | 70 | 42
  ≥1 Related TEAE leading to stopping either drug | 46 | 23

5. Secondary Outcome: Percentage of Participants With the Best Overall Response Based on the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Guidelines
Description: A best overall response rate is a CR, CRi, nPR or PR and is defined as:
  Complete Remission (CR):
  * No lymphadenopathy
  * No hepatomegaly or splenomegaly
  * Absence of constitutional symptoms
  * Polymorphonuclear leukocytes ≥ 1500/ul
  * No circulating clonal B-lymphocytes
  * Platelets > 100,000/ul
  * Hemoglobin > 11.0 g/dl
  * Normocellular <30% lymphocytes, no B-lymphoid nodules;
  Incomplete Clinical Response (CRi):
  • CR without bone marrow biopsy confirmation.
  Nodular Partial Response (nPR):
  • CR with the presence of residual clonal nodules.
  Partial Response (PR) requires:
  * ≥ 50% decrease in peripheral blood lymphocyte count
  * ≥ 50% reduction in lymphadenopathy
  * ≥ 50% reduction in size of liver and/or spleen
  * 1 or more of the following:
  * Polymorphonuclear leukocytes ≥ 1500/ul
  * Platelets >100,000/ul
Time Frame: Up to data cut-off date of 18 Feb 2013; approximately 39 months
Population: This is a smaller population used in this analysis (earlier cut-off date) prior to the last participant enrolled in the study. The Intent-to-Treat (ITT) population was defined as all participants who were randomized, independent of whether they received study treatment or not.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 212 | 215
percentage of participants | 51.9 | 62.3
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Test type: Superiority; p = 0.032, Fisher Exact; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.44 to 0.96]

6. Secondary Outcome: Percentage of Participants With a Best Overall Response Based on IWCLL Guidelines With a Later Cut-off Date of 31 March 2014
Description: A best overall response rate is a CR, CRi, nPR or PR and is defined as:
  Complete Remission (CR):
  * No lymphadenopathy
  * No hepatomegaly or splenomegaly
  * Absence of constitutional symptoms
  * Polymorphonuclear leukocytes ≥ 1500/ul
  * No circulating clonal B-lymphocytes
  * Platelets > 100,000/ul
  * Hemoglobin > 11.0 g/dl
  * Normocellular <30% lymphocytes, no B-lymphoid nodules;
  Incomplete Clinical Response (CRi):
  • CR without bone marrow biopsy confirmation.
  Nodular Partial Response:
  • CR with the presence of residual clonal nodules.
  Partial Response requires:
  * ≥ 50% decrease in peripheral blood lymphocyte count
  * ≥ 50% reduction in lymphadenopathy
  * ≥ 50% reduction in size of liver and/or spleen
  * 1 or more of the following:
  * Polymorphonuclear leukocytes ≥ 1500/ul
  * Platelets >100,000/ul
Time Frame: Up to data cut-off of 31 March 2014; approximately 53 months
Population: The Intent-to-Treat population was defined as all participants who were randomized, independent of whether they received study treatment or not
Measure: Number; unit: percentage of participants with response
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 225 | 225
percentage of participants with response | 60.9 | 70.2
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Test type: Superiority; p = 0.047, Fisher Exact; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.45 to 0.98]

7. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response
Description: Duration of response was defined as the time from first nPR, PR, CRi, or CR to PD. Duration of response was censored at the last date that the patient was known to be progression-free for: 1) participants who had not progressed at the time of analysis; 2) participants who had withdrawn consent or were lost to follow-up prior to documentation of progression
Time Frame: Up to data cut-off of 18 Feb 2013; up to approximately 39 months
Population: Intent to Treat population with an objective response as of 18 Feb 2013; includes responders
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 110 | 134
weeks | NA [131.1 to NA] — NA = The median and upper limit of the CI not estimable due to insufficient number of participants with events. | 105.3 [77.4 to 123.7]
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Test type: Superiority or Other; p = 0.826, Log Rank; Hazard Ratio (HR) = 0.94, 90% CI 2-sided [0.58 to 1.52] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

8. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response With a Later Cut-off Date of 31 March 2014
Description: Duration of response was defined as the time from first nPR, PR, CRi, or CR to PD. Duration of response was censored at the last date that the patient was known to be progression-free for: 1) patients who had not progressed at the time of analysis; 2) patients who had withdrawn consent or were lost to follow-up prior to documentation of progression
Time Frame: Up to data cut-off of 31 March 2014; up to approximately 53 months
Population: Intent to Treat population with an objective response as of 31 March 2014; includes responders.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 137 | 158
weeks | NA [149.4 to NA] — NA due to large number of censored observations. | 87.1 [77.1 to 108.7]
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Test type: Superiority; p = 0.149, Log Rank; Cox Proportional Hazard = 0.71, 90% CI 2-sided [0.48 to 1.05] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

9. Secondary Outcome: Time to Response
Description: Time to response was calculated as the time from randomization to the first nPR, PR, CRi or CR based on IWCLL guidelines
Time Frame: Up to data cut-off of 18 Feb 2013; up to approximately 39 months
Population: ITT participants with an objective response as of 18 February 2013
Measure: Median (Full Range); unit: weeks
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 110 | 134
weeks | 8.6 [3.7 to 104.3] | 8.1 [3.7 to 52.7]

10. Secondary Outcome: Time to Response for a Later Cut-off Date of 31 March 2014
Description: as for outcome 9
Time Frame: Up to data cut-off of 31 March 2014; up to approximately 53 months
Population: ITT participants who had not progressed at the time of analysis; or those who had withdrawn consent or were lost to follow-up prior to documentation of progression.
Measure: Median (Full Range); unit: weeks
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 137 | 158
weeks | 10.4 [3.7 to 136.1] | 8.1 [3.7 to 68.7]

11. Secondary Outcome: Kaplan Meier Estimate of Overall Survival
Description: Overall Survival is defined as the time between randomization and death from any cause.
Time Frame: Up to data cut off of 31 March 2014; median follow-up for all participants was 18.8 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 225 | 225
Months | NA [NA to NA] — The median had not been reached and CI not estimable because of small number of events. . | 44.0 [37.3 to NA] — Upper level CI not estimable because of small number of events
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Test type: Superiority; p = 0.883, Log Rank; Cox Proportional Hazard = 1.03, 90% CI 2-sided [0.73 to 1.46] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

12. Secondary Outcome: Kaplan Meier Estimate for Overall Survival at the Final Analysis
Description: Overall Survival is defined as the time between randomization and death from any cause. Overall survival was censored at the last date that the subject was known to be alive for participants who were alive as of the data cutoff date and for participants who were lost to follow-up before death was documented.
Time Frame: Up to the last patient last visit date of 19 May 2018; median follow-up for all participants was 46.7 months
Population: The ITT population was defined as all participants who were randomized, independent of whether they received study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 225 | 225
Months | 74.3 [58.5 to 84.4] | 70.5 [57.1 to NA] — Upper CI not estimable because of censored observations.
Statistical Analysis 1: Comparison: Lenalidomide vs Chlorambucil; Test type: Superiority or Other; p = 0.709, stratified log rank; Cox Proportional Hazard = 1.06, 90% CI 2-sided [0.83 to 1.34] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

13. Secondary Outcome: Functional Assessment of Cancer Therapy-General to Create the FACT-Leukemia (FACT-Leu) Quality of Life Instrument
Description: The FACT-Leu scale is a valid, reliable, and efficient measure of leukemia-specific health-related quality of life for acute and chronic disease. The FACT-Leu is described as including 27 items that assess 17 physical symptoms (fevers, bleeding, general pain, stomach pain, chills, night sweats, bruising, lymph node swelling, weakness, tiredness, weight loss, appetite, shortness of breath, functional ability, diarrhea, concentration, and mouth sores) and 10 emotional/social concerns (frustration with activity limitation, discouraged by illness, future planning, uncertainty, worry about illness, emotional lability, isolation, infertility concern, family worry, and worry about infections).
Time Frame: Day 1 and once every 8 weeks
Population: No data were collected for the FACT-Leu QOL assessment. Analysis was not conducted due to the discontinuation of the lenalidomide arm.
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Euro Quality of Life Five Dimension (EQ-5D) Questionnaire
Description: The standardized extended version of EQ-5D was designed for the collection of health state values using a visual analogue scale (VAS) rating scale - a vertical 20 cm visual analogue scale with the end points labeled best imaginable health state at the top and worst imaginable health state at the bottom having numeric values of 100 and 0 respectively. The participant is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
Time Frame: Day 1 and once every 8 weeks
Population: No data were collected for the EQ-5D QOL assessment. The EQ-5D analysis was not conducted due to the discontinuation of the lenalidomide arm.
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants and Types of Subsequent Anti-cancer Therapies Received Post Treatment
Description: Subsequent anti-cancer therapies administered to participants following the discontinuation of study drug (either Lenalidomide or Chlorambucil)
Time Frame: Up to the last patient last visit date of 19 May 2018; median follow-up for all participants was 46.7 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 224 | 223
participants
  Participants receiving additional CLL therapy | 125 | 120
  Participants receiving alkylating agents | 107 | 106
  Participants receiving antineoplastic aents | 93 | 86
  Participants receiving antimetabolites | 34 | 24
  Participants receiving corticosteroids | 27 | 16
  Participants receiving plant alkaloids | 22 | 11
  Participants receiving cytotoxic antibiotics | 10 | 3
  Participants receiving immunosuppressants | 3 | 2
  Participants receiving therapeutic products | 4 | 3
  Participants receiving other unspecified products | 0 | 2
  Antihistamine For Systemic Use | 1 | 1
  Drugs for Peptic ulcer and Gastric Reflex | 1 | 0
  Immunoglobulins | 1 | 2
  Other Analgesics and Antipyretics | 1 | 1
  Specific Antirheumatic Agents | 1 | 0
  Antiemetics and Antinauseants | 0 | 1
  Corticosteriods for Systemic Use | 0 | 1
  Immunostimulants | 0 | 1

16. Other Pre Specified Outcome: Number of Participants Deaths During the Treatment and Survival Follow-Up Phase
Description: The number of study participants deaths during the treatment and follow-up phase
Time Frame: From the first dose of study drug up to the last patient last visit date of 19 May 2018; median follow-up for all participants was 46.7 months
Population: ITT population includes all participants who were randomized, independent of whether they received study treatment or not
Measure: Number; unit: Participants
Arm/Group | Lenalidomide | Chlorambucil
Number analyzed (Participants) | 225 | 225
Participants | 101 | 95

ADVERSE EVENTS:
Time Frame: All AEs were recorded by the Investigator(s) from first dose of study drug to 30 days after the treatment discontinuation visit. The median treatment duration was 263 days for lenalidomide and 362 days for chlorambucil.
Description: Secondary Primary Malignancies (SPMs) were monitored and reported as SAEs regardless of the treatment arm the participant was is on. SPMs were reported from the time of signing the informed consent up to and including the survival follow-up period. Participants were followed for at least 5 years from the date the last participant was randomized.
Groups:
- Lenalidomide: For participants with normal renal function [defined as Creatinine Clearance (CrCL ) ≥ 60 mL/min], 5 mg lenalidomide was administered by mouth (PO) once daily (QD) on Days 1 through 28 of the first 28-day cycle, 10 mg lenalidomide PO QD on Days 1 through 28 starting at cycle 2, 15 mg lenalidomide PO QD starting at cycle 3 and for the remainder of the study until progressive disease (PD) or unacceptable toxicity, whichever occurred first. For participants with moderate renal impairment (defined as CrCL ≥ 30 to < 60 mL/min), 2.5 mg lenalidomide PO QD on Days 1 through 28 of the first 28-day cycle, 5 mg lenalidomide PO QD on Days 1 through 28 starting at cycle 2, 7.5 mg lenalidomide PO QD starting at cycle 3 and for the remainder of the study until PD or unacceptable toxicity, whichever occurred first.
- Chlorambucil: Chlorambucil oral tablets at 0.8 mg/kg on Days 1 and 15 of each 28-day cycle for a total duration of 12 months
Arm/Group | Lenalidomide | Chlorambucil
All-Cause Mortality (participants affected / at risk) | 100/224 | 93/223
Serious Adverse Events (participants affected / at risk) | 148/224 | 90/223
Other Adverse Events (participants affected / at risk) | 204/224 | 184/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=224) | Chlorambucil (N=223)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 18 | 10
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 3 | 4
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 3
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 54 | 33
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
SPLENIC HAEMORRHAGE (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 19 | 13
ANGINA PECTORIS (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 4 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 4 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 3 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 2 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
DIPLOPIA (Eye disorders) | 0 | 1
MACULOPATHY (Eye disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2
COLITIS (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
FEMORAL HERNIA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 2
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 3
ASTHENIA (General disorders) | 0 | 3
FATIGUE (General disorders) | 2 | 2
MULTI-ORGAN FAILURE (General disorders) | 3 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PAIN (General disorders) | 0 | 1
PYREXIA (General disorders) | 10 | 6
SUDDEN CARDIAC DEATH (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 2
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 1
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 2 | 1
CELLULITIS (Infections and infestations) | 2 | 3
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0
ENTEROBACTER SEPSIS (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 1 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1
LUNG INFECTION (Infections and infestations) | 2 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
PELVIC INFECTION (Infections and infestations) | 1 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 24 | 6
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 4
SEPSIS SYNDROME (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1
BLOOD UREA INCREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 3
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2
GOUT (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 3
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 2 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8
BASOSQUAMOUS CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RICHTER'S SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
SQUAMOUS CELL CARCINOMA OF THE ORAL CAVITY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 1
SIMPLE PARTIAL SEIZURES (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 3 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 2 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 4 | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
LERICHE SYNDROME (Vascular disorders) | 1 | 0
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 | 0
SHOCK (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=224) | Chlorambucil (N=223)
NEUTROPENIA (Blood and lymphatic system disorders) | 126 | 74
VOMITING (Gastrointestinal disorders) | 11 | 28
ASTHENIA (General disorders) | 19 | 10
PYREXIA (General disorders) | 37 | 18
NASOPHARYNGITIS (Infections and infestations) | 12 | 3
PNEUMONIA (Infections and infestations) | 13 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 30 | 13
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 16 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 | 12
ANAEMIA (Blood and lymphatic system disorders) | 69 | 46
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 72 | 50
ABDOMINAL PAIN (Gastrointestinal disorders) | 30 | 10
CONSTIPATION (Gastrointestinal disorders) | 28 | 17
DIARRHOEA (Gastrointestinal disorders) | 66 | 32
NAUSEA (Gastrointestinal disorders) | 33 | 63
FATIGUE (General disorders) | 66 | 53
OEDEMA PERIPHERAL (General disorders) | 43 | 16
BRONCHITIS (Infections and infestations) | 16 | 4
INFLUENZA (Infections and infestations) | 13 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 | 11
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 14 | 7
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 14 | 7
BLOOD CREATININE INCREASED (Investigations) | 22 | 7
WEIGHT DECREASED (Investigations) | 34 | 23
HYPERKALAEMIA (Metabolism and nutrition disorders) | 12 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 12
BACK PAIN (Musculoskeletal and connective tissue disorders) | 28 | 18
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 15 | 5
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 85 | 11
DIZZINESS (Nervous system disorders) | 16 | 12
HEADACHE (Nervous system disorders) | 16 | 11
INSOMNIA (Psychiatric disorders) | 14 | 11
COUGH (Respiratory, thoracic and mediastinal disorders) | 38 | 21
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 24 | 14
PRURITUS (Skin and subcutaneous tissue disorders) | 18 | 7
RASH (Skin and subcutaneous tissue disorders) | 41 | 19

LIMITATIONS AND CAVEATS:
After notification by the US Food and Drug Administration on 12Jul2013, Celgene agreed to stop lenalidomide due to an imbalance in the number of deaths on the lenalidomide arm versus the chlorambucil arm; no causality for the imbalance was identified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 12 months since study completion. Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.